CLINICAL TRIAL: NCT00055822
Title: A Phase I/II Study of Oblimersen Sodium (G3139, Genasense) in Combination With Oxaliplatin, 5FU and Leucovorin (FOLFOX4) Regimen in Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy and Oblimersen in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271308; U01CA069853 (NIH); P30CA054174 (NIH); SACI-IDD-02-23 (Other: San Antonio Cancer Institute); NCI-5793 (Other: NCI)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — oblimersen; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: oblimersen sodium
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Oblimersen may increase the effectiveness of chemotherapy by making tumor cells more sensitive to the drugs.

PURPOSE: Phase I/II trial to study the effectiveness of combining oxaliplatin, fluorouracil, and leucovorin with oblimersen in treating patients who have unresectable, metastatic, or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oblimersen when administered with oxaliplatin, fluorouracil, and leucovorin calcium in patients with advanced colorectal cancer.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.
* Determine the plasma pharmacokinetics of oblimersen and oxaliplatin in patients treated with this regimen.
* Determine relevant predictive biomarkers of response in patients treated with this regimen.

OUTLINE: This is an open-label, phase I, dose-escalation study of oblimersen followed by a non-randomized, phase II study.

* Phase I: Patients receive oblimersen IV continuously on days 1-5 and 15-19; leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 6, 7, 20, and 21; and oxaliplatin IV over 2 hours on days 6 and 20.

Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

* Phase II: Up to 35 additional patients are treated as in phase I, with oblimersen at the MTD.

In both phases, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 6-53 patients (6-18 patients for phase I and 12-35 patients for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum

  * Unresectable, metastatic, or recurrent disease
* Measurable or evaluable disease (phase I)
* Measurable disease (phase II)
* No known brain metastases

  * Patients with previously treated brain metastases who are not currently receiving steroids and have a stable CT scan or MRI are eligible

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* INR no greater than 1.5 times ULN (unless currently receiving anticoagulant therapy)
* PT/PTT no greater than 1.5 times ULN (unless currently receiving anticoagulant therapy)

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction to compounds of similar chemical or biologic composition to fluorouracil or oxaliplatin
* No other concurrent uncontrolled medical condition that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No known history of degenerative facet disease during prior fluorouracil therapy
* No HIV-positive patients receiving combination antiretroviral therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent epoetin alfa during course 1
* No concurrent routine filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent immunotherapy

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No prior oblimersen
* No other concurrent investigational agents
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, MD, Study Chair — San Antonio Cancer Institute
Locations (1):
- San Antonio Cancer Institute, San Antonio, Texas, United States